CLINICAL TRIAL: NCT02890186
Title: Dual-loop Target Controlled Infusion for Coadministration of Propofol and Remifentanil Guided by Narcotrend Index in Anterior Cervical Decompression and Fusion With Internal Fixation
Brief Title: Dual-loop Target Controlled Infusion for Coadministration of Propofol and Remifentanil Guided by Narcotrend Index
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Guangzhou General Hospital of Guangzhou Military Command (Other)
Responsible Party: Principal Investigator, bo xu, associate chief physician, Guangzhou General Hospital of Guangzhou Military Command
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: double closed-loop
Record Dates: First submitted 2016-08-16; First posted 2016-09-07 (Estimated); Last update posted 2016-09-07 (Estimated); Status verified 2016-08

CONDITIONS: Anesthesia
Keywords: narcotrend; propofol; remifentanil; closed-loop of target controlled infusion
MeSH Terms: interventions — Ecological Momentary Assessment

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Dual-Loop TCI (Experimental): the investigator modified the effect-site target concentrations by NI.If NI fall down to 46 and keep 46 more than 30 seconds,propofol and remifentanil were infused as feedback automatically to achieve the target NI of 26-46.
  Interventions: Device: Narcotrend
- manual (Placebo Comparator): the investigator modified the effect-site target concentrations of both drugs without minimum or maximum concentration limits without using the Narcotrend monitor only depend on the experience of anesthesiologist.
  Interventions: Other: experience

INTERVENTIONS:
Device: Narcotrend — the investigator modified the effect-site target concentrations by NI.If NI fall down to 46 and keep 46 more than 30 seconds,propofol and remifentanil were infused as feedback automatically to achieve the target NI of 26-46.
  Other Names: Dual-Loop Target Controlled Infusion of Propofol and Remifentanil Guided by Narcotrend Index
  Arms: Dual-Loop TCI
Other: experience — the investigator modified the effect-site target concentrations of both drugs without minimum or maximum concentration limits without using the Narcotrend monitor only depend on the experience of anesthesiologist.
  Other Names: Control infusion of propofol and remifentanil guided by experience
  Arms: manual

SUMMARY:
To investigate the application of closed target-controlled infusion(TCI) of propofol and remifentanil guided by Narcotrend index in the anterior cervical decompression and fusion with internal fixation surgery.

DETAILED DESCRIPTION:
Sixty patients scheduled for anterior cervical decompression and fusion with internal fixation surgery under general anesthesia were randomly divided into two groups:closed-loop (group A,n=30) and open-loop group(group B,n=30).The procedure during induction of anesthesia was same in two groups.In group A,if Narcotrend index(NI) fall down to 46 and keep more than 30 seconds,propofol and remifentanil were intravenously infused as feedback automatically to achieve the target NI of 26-46.However,the NI in group B was controlled manually.

ELIGIBILITY:
Inclusion Criteria:

1. ASA Ⅰ ~ Ⅱ women undergoing Laparoscopic surgery.
2. Written informed consent from the patient or the relatives of the participating patient.
3. BMI:18.0～25 kg/m2

Exclusion Criteria:

1. Mental illness can not match
2. epidural anesthesia contraindicated
3. People who have Slow-type arrhythmias
4. Chronic renal failure
5. Alcohol or drug abuse
6. Already taking gabapentin, pregabalin, benzodiazepin or antidepression drug

Ages: 23 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2016-04; Primary Completion 2016-09 (Estimated); Study Completion 2016-09 (Estimated)

PRIMARY OUTCOMES:
the total dose of propofol and remifentanil | within three hours from the beginning to the end of the propofol and remifentanil
  record the total dose of propofol and remifentanil from the beginning to the end of anesthesia

CONTACTS AND LOCATIONS:
Locations (1):
- Guangzhou Military Region General Hospital, Department of Anesthesiology, Guangzhou, Guangdong, China